CLINICAL TRIAL: NCT04430101
Title: Stability and Outcomes of Non-displaced Lisfranc Injuries - A Prospective Multicenter Cohort Study
Brief Title: Stability and Outcomes of Non-displaced Lisfranc Injuries
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20/00913
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Lisfranc Injury; Sprain of Foot
Keywords: Lisfranc injury; Weightbearing radiographs; Stress fluoroscopy; Homerun screw
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Participants are evaluated by weightbearing radiographs. Patients with no signs of dislocation on the weightbearing radiographs will undergo stress fluoroscopy. Patients with negative stress fluoroscopy are allocated to Cohort 1, patients with positive stress fluoroscopy are allocated to Cohort 2.
  The study design is a non-inferiority study, proving to show that the outcomes of Cohort 2 are non-inferior compared to Cohort 1.
  Patients with positive weightbearing radiographs (interval between medial cuneiform and base of second metatarsal increased by > 2 mm compared to the contralateral side) will be operated with minimally invasive stabilization (eg. isolated "homerun screw") and followed up prospectively as a single cohort (Cohort 3).
Who Masked: Participant
Masking Description: The participants will be blinded for the result of the stress fluoroscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Negative WB radiographs and stress fluoroscopy (Active Comparator): Cohort 1
  Negative weight bearing radiographs:
  Interval between medial cuneiform and base of the second metatarsal (C1-M2) are less than 2mm increased compared to the uninjured side.
  Negative stress fluoroscopy: the midfoot is tested stable
  Interventions: Procedure: Conservative treatment
- Negative WB radiographs / positive stress fluoroscopy (Active Comparator): Cohort 2
  Negative weight bearing radiographs:
  Interval between medial cuneiform and base of the second metatarsal (C1-M2) are less than 2mm increased compared to the uninjured side.
  Positive stress fluoroscopy: manual testing reveals midfoot instability
  Interventions: Procedure: Conservative treatment
- Surgical cohort (Cohort 3) (Other): Patients with positive weightbearing radiographs will be operated on with minimally invasive technique and followed up as an independent cohort.
  Interventions: Procedure: Minimally invasive stabilization of Lisfranc injuries

INTERVENTIONS:
Procedure: Minimally invasive stabilization of Lisfranc injuries — Patients with positive weightbearing radiographs will be operated by minimally invasive stabilization (eg, isolated homerun screw)
  Arms: Surgical cohort (Cohort 3)
Procedure: Conservative treatment — Patients with negative weightbearing radiographs will be treated conservatively
  Arms: Negative WB radiographs / positive stress fluoroscopy; Negative WB radiographs and stress fluoroscopy

SUMMARY:
In this multicenter cohort study, the stability of non-displaced Lisfranc injuries as well as their outcomes will be evaluated.

DETAILED DESCRIPTION:
Injuries to the tarsometatarsal joints ("Lisfranc injuries") that are non-displaced on non-weightbearing radiographs and CT are common injuries. To refer these injuries to the right treatment, evaluating their stability is essential. For this purpose, both weightbearing radiographs and stress fluoroscopy have been proposed. However, there is no consensus concerning both the use and interpretation of weightbearing radiographs and no standardized technique and interpretation of stress fluoroscopy in non-displaced Lisfranc injuries.

In the current study, participants will be assigned to non-operative or operative treatment based on Lisfranc joint stability evaluation by weightbearing radiographs.

All Patients with negative weightbearing radiographs will be treated conservatively. In addition, their injured feet will be evaluated by manual stress fluoroscopy. Depending on the result of the stress fluoroscopy (positive/negative), the conservatively treated patients will be assigned to 2 cohorts, whose outcomes will be compared.

Patients with positive weightbearing radiographs will be treated operatively by minimally invasive stabilization of the midfoot (eg. isolated "homerun screw"). The operatively treated patients will be followed up as an independent cohort.

ELIGIBILITY:
Inclusion Criteria:

* Acute Lisfranc injuries that are non-displaced (< 2mm) on non-weightbearing radiographs and CT
* Patients between 18 and 70 years of age
* Acute presentation at one of our departments, enabling evaluating the stability of the injuries within 4 weeks

Exclusion Criteria:

* Fractures with an intraarticular step of > 2mm on the initial non weight-bearing radiographs and/or CT
* Delayed presentation (weight-bearing radiographs taken > 4 weeks after injury)
* Bilateral injuries
* Concomitant major injuries of the foot, ankle or leg that affect the rehabilitation process
* Multitraumized patients
* Previous injury or surgery of the mid foot
* Charcot foot
* Noncompliant patients
* Insufficient Norwegian or English language skills
* Patients not available for follow-up
* Inability to conduct the rehabilitation protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Manchester-Oxford Foot Questionnaire (MOxFQ) | 5 years
  Foot-Ankle specific PROM (0-100 with 0 representing the best possible outcome)

SECONDARY OUTCOMES:
American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Midfoot score | 5 years
  Widely used foot/ankle score (0-100 with 100 representing the best possible outcome)
Self-reported foot and ankle score (SEFAS) | 5 years
  Foot-Ankle specific PROM (0-48 with 48 representing the best possible outcome)
Visual Analogue Scale (VAS) for pain | 5 years
  Scores pain at rest and on activity (0-10 with 0 representing no pain)
Short-Form (SF) 36 | 5 years
  Patient reported score measuring quality of life and health status
Posttraumatic osteoarthritis | 5 years
  The presence of osteoarthritis of the tarsometatarsal joints is graded based on the Brodén radiographs taken at 1 year, 2 year and 5 year follow-up using the Kellgren & Lawrence classification system.
Incidence of complications | 5 years
  Yes/no for deep or superficial infection, nerve or tendon injury, deep venous thrombosis, hardware complaints and secondary surgery. Regards the patients that have undergone surgical treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Molund, MD, Principal Investigator — Ostfold Hospital Trust
Locations (2):
- Norway (2):
  - Oslo university hospial, Oslo
  - Østfold Hospital Trust, Sarpsborg, Østfold fylke

IPD SHARING:
Plan to Share IPD: No